CLINICAL TRIAL: NCT05019963
Title: Enhancing COVID Rehabilitation With Technology (ECORT): An Open-label, Single Site Randomized Controlled Trial Evaluating the Effectiveness of Electronic Case Management for Individuals With Persistent COVID-19 Symptoms.
Brief Title: Enhancing COVID Rehabilitation With Technology
Acronym: ECORT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Simon Hatcher, Acting Chair, Department of Psychiatry, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210533-01H
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Covid19
Keywords: Long COVID; Post-COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Assessment. Participants randomized to the control arm will be offered assessment by a clinician, guided by the WHO Post COVID-19 case report form. This is a clinical tool developed by WHO to guide and document the sequelae of COVID-19 and to ensure that clinical and rehabilitation needs are identified.
  Investigation. Clinician judgement will be used to decide on further testing needed for clinical care.
  Management. Control participants will receive a rehabilitation plan developed with their health professional that will be implemented in the eight weeks after their initial consultation (baseline visit). The implementation will involve face to face or virtual care from a registered health professional provided by the clinic or research staff. This may be a combination of, but not limited to, occupational therapy, physical therapy and/or social work/counselling. The frequency of treatment visits will depend on the individual treatment plan after assessment.
  Interventions: Other: Usual Care
- Electronic Case Management plus Usual Care (Experimental): Participants randomized to the experimental arm will receive assessment, investigation and management as the Active Comparator Arm plus access to an electronic case management platform - NexJ Connected Wellness (https://nexjhealth.com/) which complements the rehabilitation plan. This would include for example setting targets for activity that would be monitored with NexJ; educational materials; and support with medication adherence by reminders. The NexJ platform will include the following sections: Trusted Educational Content (Health Library); Symptom Tracking, Goal Setting, Community Forums and Reporting.
  Interventions: Behavioral: NexJ Connected Wellness; Other: Usual Care

INTERVENTIONS:
Behavioral: NexJ Connected Wellness — NexJ Connected Wellness is an electronic case management platform with a patient-facing smart phone application and a clinician-facing web dashboard.
  Arms: Electronic Case Management plus Usual Care
Other: Usual Care — Participants will receive a treatment plan as decided on with their clinician(s).

SUMMARY:
In March 2020, the World Health Organization (WHO) declared the novel coronavirus (COVID-19) a global pandemic. Ontario has confirmed more than 547,000 cases of COVID-19 since testing began. For many of these patients, symptoms resolve within 4 weeks of onset. However, it is becoming apparent that a significant number of individuals are experiencing symptoms that persist long after the acute infection, known as Long COVID. These individuals have a wide constellation of presenting symptoms, often varying from initial presentation. For this study, we will be enrolling individuals receiving care at The Ottawa Hospital for Long COVID. This study aims to determine the following four things: 1) will adding electronic case management improve quality of life three months after coming to hospital with Long COVID; 2) is the electronic case management platform cost effective; 3) is there any factors that predict outcomes at 3 months; 4) to determine how a personalized rehabilitation program supported by a digital platform could be implemented for individuals with Long COVID. We will enroll individuals from The Ottawa Hospital who will then be randomly assigned to receive either usual care or usual care plus electronic case management, through a platform called NexJ Connected Wellness. Participants will also complete questionnaires every 4 weeks for 3 months. We will be looking at quality of life, mental and physical health, cognitive symptoms, fatigue and pain.

ELIGIBILITY:
Inclusion Criteria

Participants must:

1. Be 18 years of age or older
2. Have a confirmed diagnosis of COVID-19 with a PCR test at least 12 weeks prior OR a confirmed Rapid Antigen Test at least 12-weeks prior OR meet Ottawa Public Health guidance for a suspected COVID-19 case
3. Have at least one ongoing symptom consistent with Long COVID as measured by the WHO Post COVID Case Report Form (CRF)
4. Have a minimum WHODAS (36 item) sum score of 15
5. Be willing to use email for study activities
6. Be able and willing to use a smart phone application for the duration of the trial
7. Be able to read and understand English or French.
8. Be willing and able to provide informed consent.

Exclusion Criteria

Participants must not:

1. Have any significant functional impairment (for example. advanced dementia, heart or lung disease) as judged by the assessing clinician
2. Participate in another long-COVID trial where treatment is required in the protocol (pharmacological or behavioural). Observational studies will be allowed.
3. Have symptoms consistent with Long COVID that are better explained by an alternative diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in WHODAS 2.0 score | Baseline and Week 12
  The WHODAS is the 36-item self report questionnaire measuring health and disability from the previous 30 days across six domains of functioning: cognition, mobility, self-care, getting along, life activities and participation. Responses are scored on a 5 point Likert scale: None (0), Mild (1), Moderate (2), Severe (3), and Extreme/Cannot Do (4). Change from baseline to week 12 will be measured as primary outcome.

SECONDARY OUTCOMES:
WHO Post-COVID CRF | Module 1 will be administered at baseline only. Modules 2 and 3 will be administered at baseline and 12 weeks.
  The WHO Post-COVID CRF will measure characteristics of COVID-19 infection and post-COVID symptoms including demographics, pregnancy, pre-COVID health status, and details about the acute COVID infection, vaccination status, occupational status, functioning, post-COVID symptoms, clinical tests and scales (including neurological, radiographic, blood tests, heart and lung function, mental health, function, and musculoskeletal tests) new diagnoses or complications related to COVID infection, and health service use, symptoms.
PHQ-9 | Baseline, Week 4, Week8 and Week 12
  A 9-item questionnaire that assesses the severity of depression symptoms experienced within the last two weeks. Participants are asked to rate each symptom of depression on a Likert scale from 0 (not at all) to 3 (nearly every day).
GAD-7 | Baseline, Week 4, Week8 and Week 12
  A 7-item questionnaire that assesses the severity of anxiety symptoms experienced within the last two weeks.
PSQI | Baseline, Week 4, Week8 and Week 12
  The Pittsburgh Sleep Quality Index is a self-report questionnaire that assesses sleep quality in the previous month and takes 5-10 minutes to complete. It has been translated into over 50 languages.
PCL-5 | Baseline, Week 4, Week8 and Week 12
  A 20-item self-report measure that assesses the presence and severity of PTSD symptoms, corresponding with DSM-5 criteria for PTSD
EQ-5D-5L | Baseline, Week 4, Week8 and Week 12
  This is a 5-item questionnaire that assesses health-related quality of life, including mobility, self-care, ability to participate in one's usual activities, pain or discomfort, and anxiety or depression and a Visual Analogue Scale (VAS) which asks participants to evaluate their overall health on a scale from 0-100.
Fatigue Severity Scale | Baseline, Week 4, Week8 and Week 12
  The Fatigue Severity Scale is a 9-item self-report that measures the severity and functional impact of fatigue.
Fatigue Numeric Rating Scale | Baseline, Week 4, Week8 and Week 12
  A single item patient reported outcome, scored on a scale of 0-10.
Pain Numeric Rating Scale | Baseline, Week 4, Week8 and Week 12
  The Pain Numeric Rating Scale will be used to assess pain intensity using a 0-10 ranking scale, where 0 represents "no pain" and 10 "unbearable pain".
MRC Dyspnoea Scale | Baseline, Week 4, Week8 and Week 12
  A 5-item self report scale that evaluates statements of perceived breathlessness.
WEMWBS | Baseline and Week 12
  The Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) (short version) is a 7-item scale which measures multiple aspects of mental wellbeing.
Oral Trail Making Test A and B | Baseline and Week 12
  Used to evaluate executive function, visual attention and task switching in participants. During TMT A, participants will be asked to count down out louad as quickly as they can sequentially, starting at "1" until the end. During TMT B, participants will be asked to speak outloud, alternating between numbers and letters (e.g. 1-A-2-B etc).
Hopkins Verbal Learning Test-Revised (HVLT-R) | Baseline and Week 12
  The Hopkins Verbal Learning Test-Revised (HVLT-R) will be used to evaluate verbal learning and memory capabilities in participants33. The HVLT consists of a 12-item word list, composed of four words from each of three semantic categories.
Digit Span subset | Baseline and Week 12
  The Digit Span subset, a component of the Working Memory Index of the Weschler's Adult Intelligence Scale - 4th Edition (WAIS-IV), will be used to assess attention and working memory34. Participants will be read a series of numbers and then asked to recall the numbers to the examiner in order (forward span), in reverse order (backward span) and in sequence (sequence span).
Phonemic and Semantic Verbal Fluency (or Controlled Oral Word Association Test) | Baseline and Week 12
  The Phonemic and Semantic Verbal Fluency (or Controlled Oral Word Association Test) test will be used to assess verbal fluency. Participants will be given one minute to produce as many unique words as possible: 1) within a semantic category (category fluency for Animals); and 2) starting with a given letter (letter fluency for letters F, A and S).
AUDIT | Baseline
  Alcohol use: The AUDIT questionnaire is designed to assess alcohol consumption, drinking behavior, adverse reactions, alcohol-related problems. Among those who were known to misuse alcohol, the AUDIT successfully detected an alcohol use disorder 99% of the time 53. The AUDIT-C is the first 3-items of the AUDIT and will be used as a screening questionnaire. Participants who score above 4 on the AUDIT-C will also be asked to complete the Full AUDIT (the additional seven questions).
ASSIST | Baseline
  Alcohol and Substance Use: The ASSIST is a clinical interview collecting information regarding use of tobacco, alcohol, cannabis, cocaine, amphetamine type stimulants, sedatives, hallucinogens, inhalants, opioids, and other drugs. Internal Consistency (Chronbach's alpha) was over 0.80 for the majority of domains and good concurrent validity

CONTACTS AND LOCATIONS:
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The Principal Investigator will retain ownership of the dataset through the 10 year archiving period. The protocol will be published, at a minimum on an open-science platform (e.g. Open Science Framework or medRXiv). If the protocol is published in an academic journal, the Principal Investigator will ensure it is open access. The anonymized data set will be shared on an open access platform, such as Open Science Framework or Zenodo. The anonymized dataset may also be shared with the WHO to facilitate global post-COVID-19 research and treatment efforts.
Supporting Information: Study Protocol, ICF
Time Frame: The study protocol will become available as soon as possible after ethical approval and implementation. The informed consent form will be shared as supporting documentation with the protocol.

REFERENCES:
- [Derived] Hatcher S, Werier J, Edgar NE, Booth J, Cameron DWJ, Corrales-Medina V, Corsi D, Cowan J, Giguere P, Kaluzienski M, Marshall S, Mestre T, Mulligan B, Orpana H, Pontefract A, Stafford D, Thavorn K, Trudel G. Enhancing COVID Rehabilitation with Technology (ECORT): protocol for an open-label, single-site randomized controlled trial evaluating the effectiveness of electronic case management for individuals with persistent COVID-19 symptoms. Trials. 2022 Sep 2;23(1):728. doi: 10.1186/s13063-022-06578-1. PMID 36056372